CLINICAL TRIAL: NCT03416283
Title: Remote Monitoring and Enhanced Social Support for Hypertension Management
Brief Title: Remote Monitoring and Social Support for Hypertension Management
Acronym: SupportBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 828417
Record Dates: First submitted 2018-01-17; First posted 2018-01-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Remote Patient Monitoring

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote Monitoring (RM) (Experimental): Remote Monitoring subjects will receive a blood pressure cuff and bidirectional text messaging regarding blood pressure and medication adherence.
  Interventions: Behavioral: Remote Monitoring
- Remote Monitoring + Social Support (RM+SS) (Experimental): Remote Monitoring + Social Support subjects will receive a blood pressure cuff and bidirectional text messaging regarding blood pressure and medication adherence, as well as a social support partner to provide additional feedback to the participant on their monitoring and adherence practices.
  Interventions: Behavioral: Remote Monitoring + Social Support
- Usual Care (No Intervention): Usual care subjects will not receive a blood pressure cuff or bidirectional text messaging. They will be asked to take their medication and monitor BP as usual with no additional contact from study staff until the 4 month study follow-up.

INTERVENTIONS:
Behavioral: Remote Monitoring — Remote BP monitoring and medication adherence
  Arms: Remote Monitoring (RM)
Behavioral: Remote Monitoring + Social Support — Remote BP monitoring and medication adherence with enhanced support from a support partner ("facilitated cheerleading")
  Arms: Remote Monitoring + Social Support (RM+SS)

SUMMARY:
A 3-arm randomized pilot trial aimed at comparing the effectiveness of different remote approaches to improving blood pressure (BP) control.

DETAILED DESCRIPTION:
The investigators plan to leverage the Way to Health (WTH) platform to develop and evaluate a new HTN service-delivery model that is integrated with routine clinical care at Penn Family Care (PFC), an academic family medicine practice in West Philadelphia. Among patients with poorly controlled HTN:

1. The investigators will assess the effects of monitoring blood pressure and medication adherence with feedback to the patient and to the clinical practice, as needed if out of control.
2. The investigators will also compare the impact of providing feedback to a social support partner with facilitated cheerleading.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years old with HTN (ICD-10 code I10)
* Has had at least two office visits at Penn Family Care (PFC) within the past 12 months (at time of chart review), with at least two of the visits with BP readings exceeding HTN guidelines, including the last visit (150/90 or 140/90 if ages 21-59 yrs with CKD or diabetes)
* Must have a cellular phone with texting capabilities
* Must be prescribed at least one medication for hypertension

Exclusion Criteria:

* Has metastatic (Stage IV) blood or solid tumor cancer
* Has end stage renal disease
* Has congestive heart failure
* Has dementia
* Has liver cirrhosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-10-26 (Actual); Study Completion 2019-10-26 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 4 months
  Systolic blood pressure during the 4-month study visit, adjusted for initial systolic blood pressure

SECONDARY OUTCOMES:
Percent of patients that are normotensive | 4 months
  The percent of patients with final blood pressure within the normal range.
Medication adherence | 4 months
  Medication adherence as measured by the text message response
Diastolic blood pressure | 4 months
  Adjusted for initial diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Volpp KG, Troxel AB, Teel J, Reitz CR, Purcell A, Shen H, McNelis K, Snider CK, Asch DA. Remote Blood Pressure Monitoring With Social Support for Patients With Hypertension: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2413515. doi: 10.1001/jamanetworkopen.2024.13515. PMID 38829618